CLINICAL TRIAL: NCT01863147
Title: Sitagliptin Reduces Left Ventricular Mass in Normotensive Type 2 Diabetic Patients With Coronary Artery Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wuhan General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, Xiang Guang-da, director, Wuhan General Hospital of Guangzhou Military Command
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010Wze052
Record Dates: First submitted 2013-05-21; First posted 2013-05-27 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Newly Diagnosed Type 2 Diabetes; Coronary Artery Disease
Keywords: Type 2 diabetes; left ventricular mass; inhibitor of dipeptidyl peptidase-4
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Acarbose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sitagliptin (Experimental): Sitagliptin 0.1 daily for 1 year
  Interventions: Drug: Sitagliptin and acarbose
- acarbose (Active Comparator): acarbose 150mg daily for 1 year
  Interventions: Drug: Sitagliptin and acarbose

INTERVENTIONS:
Drug: Sitagliptin and acarbose — Sitagliptin group: The intervention drug is sitagliptin. Acarbose group: The intervention drug is acarbose.

SUMMARY:
Cardiovascular complications account for the highest mortality in type 2 diabetic patients, mainly due to coronary artery disease (CAD).Left ventricular hypertrophy (LVH) is widespread in type 2 diabetic patients with CAD, even in the absence of hypertension .It is a strong predictor of cardiovascular events and all-cause mortality .

Sitagliptin, an inhibitor of dipeptidyl peptidase-4 (DPP-4), may regress left ventricular mass (LVM) in newly diagnosed type 2 diabetic patients with CAD .

ELIGIBILITY:
Inclusion Criteria:Patients had to have the levels of hemoglobin A1c (HbA1c) > 7.0 %. They also had to have either angiographically documented coronary artery disease or a previous history of myocardial infarction. In addition, they were also required to have an office BP < 135/85 mm Hg and the presence of LVH on echocardiography (American Society of Echocardiography criteria LVM index [LVMI] > 115 g/m2 for men and > 95 g/m2 for women) . -

Exclusion Criteria:Patients were excluded if they were currently prescribed glucagon-like peptide (GLP) -1 analogues or DPP-4 inhibitors or glucosidase inhibitor or anti-hypertensive drugs (including b-blockers), diabetes medications, estrogen supplements, thyroxine, diuretics, hypolipidemic drugs. They were also excluded if they had renal and liver dysfunction, heart failure, or malignancy, or were unable to give informed consent. Patients with contraindications to cardiac magnetic resonance (CMR) (pacemakers, claustrophobia) were also excluded, as were pregnant or lactating women. -

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Left ventricular mass and left ventricular volume | 2013~2014(follow up 1 year)
  Cardiac magnetic resonance (CMR) imaging was performed at baseline and at 12 months for left ventricular mass and left ventricular volume.

SECONDARY OUTCOMES:
Endothelial function and augmentation index (AIx) | 2013~2014 (follow up 1 year)
  1. Endothelial function was assessed on three visits (baseline, month 6, and month 12) by measuring flow-mediated dilation (FMD) of the brachial artery in response to hyperemia according to our previous reports.
  2. Pulse wave analysis and pulse wave velocity (PWV) were measured at baseline, 6 months visit, and 12 months visit.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Guangda, MD,PhD, Study Director — Wuhan General Hospital of Guangzhou Command
Locations (2):
- China (2):
  - Guangda Xiang, Wuhan, Hubei
  - Wuhan General Hospital, Wuhan, Hubei